CLINICAL TRIAL: NCT04039659
Title: POstoperative Negative-pressure Incision Therapy Following LIver TRANSplant (PONILITRANS Study): a Randomized Controlled Trial
Brief Title: POstoperative Negative-pressure Incision Therapy Following LIver TRANSplant:a Randomized Controlled Trial
Acronym: PONILITRANS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitario Virgen de la Arrixaca (Other)
Responsible Party: Principal Investigator, Ana Delegido Garcia, Principal investigator, Hospital Universitario Virgen de la Arrixaca
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2019-1-6-HCUVA
Record Dates: First submitted 2019-06-10; First posted 2019-07-31 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Liver Transplant; Complications
Keywords: wound complications; negative-pressure wound therapy
MeSH Terms: interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Intervention Model Description: After signing the informed consent of those patients who meet the inclusion criteria, they will be randomized into two groups to install the PICOⓇ device or conventional dressings over the wound. After 7 days, the PICOⓇ device will be removed and both preoperative and postoperative variables will be studied.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (No Intervention): Patients will be cured with dressings wound everyday or before if there are complications in surgical incisions.
- PICO group (Active Comparator): Patients will carry the device for 7 days uninterrupted until its withdrawal.
  Interventions: Device: Negative-pressure wound therapy (PICO)

INTERVENTIONS:
Device: Negative-pressure wound therapy (PICO) — After the selection of patients and the signing of the consent, patients will be randomized and the device will be placed to those who belong to the PICO group in the operating room.
  Arms: PICO group

SUMMARY:
This study is to evaluate whether the prophylactic use of a negativa pressure therapy device (PICOⓇ) on the closed wound of the liver transplant, reduces the postoperative complications of surgical wounds, compared to the use of dressings conventional postoperative

DETAILED DESCRIPTION:
Postoperative complications of surgical wounds are frequent after surgical procedures, even more in the context of liver transplantation given the necessary immunosuppression, high surgical time, high hospital stay and intensive care, politransfusions, etc. Negative pressure therapy is well established for the treatment of open wounds, its use having been recently indicated on closed surgical wounds. The evidence to justify this intervention is still limited.

The objective of our clinical trial is to evaluate whether the prophylactic use of a negative pressure therapy device (PICOⓇ) on the closed wound of the liver transplant, reduces the postoperative complications of surgical wounds, compared to the use of dressings conventional postoperative After signing the informed consent of those patients who meet the inclusion criteria, they will be randomized into two groups to install the PICOⓇ device or conventional dressings on the wound. After 7 days, the PICOⓇ device will be removed and both preoperative and postoperative variables will be studied in terms of incidence of surgical site events, stay, etc.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes aged between 18 and 70 years included in the waiting list for liver transplantation by the committee of the Virgen de la Arrixaca University Hospital.

Exclusion Criteria:

* To have been rejected for liver transplantation by said committee

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of surgical site | 30 days after surgery
  Any complication of surgical site will be registered

SECONDARY OUTCOMES:
Quality of life of transplantation patient | 6 months
  We will use Cardiff Wound Impact Schedule to evaluate the possible improvement in the quality of life of transplantation patients derived from the decrease in the requirement of health resources.
Nosocomial infection rate | 30 days after surgery (3rd, 7th, 15th and 30th post trasplant)
  To verify the change in rates of nosocomial infections in the context of liver transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Delegido García, Principal Investigator — Hospital Universitario Virgen de la Arrixaca
Locations (1):
- Hospital Clínico Universitario Virgen de la Arrixaca, El Palmar, Murcia, Spain

IPD SHARING:
Plan to Share IPD: Yes
All documentation related to the study will remain stored in the Investigator's Archive, in the participating center, in the custody of the Principal Investigator until the end of it. Once the study is finished, the documentation will be indexed and will go to the general file of the center.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available when the results are published.

REFERENCES:
- [Background] Culver DH, Horan TC, Gaynes RP, Martone WJ, Jarvis WR, Emori TG, Banerjee SN, Edwards JR, Tolson JS, Henderson TS, et al. Surgical wound infection rates by wound class, operative procedure, and patient risk index. National Nosocomial Infections Surveillance System. Am J Med. 1991 Sep 16;91(3B):152S-157S. doi: 10.1016/0002-9343(91)90361-z. PMID 1656747
- [Background] Haley RW, Culver DH, Morgan WM, White JW, Emori TG, Hooton TM. Identifying patients at high risk of surgical wound infection. A simple multivariate index of patient susceptibility and wound contamination. Am J Epidemiol. 1985 Feb;121(2):206-15. doi: 10.1093/oxfordjournals.aje.a113991. PMID 4014116
- [Background] Webster J, Scuffham P, Sherriff KL, Stankiewicz M, Chaboyer WP. Negative pressure wound therapy for skin grafts and surgical wounds healing by primary intention. Cochrane Database Syst Rev. 2012 Apr 18;(4):CD009261. doi: 10.1002/14651858.CD009261.pub2. PMID 22513974
- [Background] Kilpadi DV, Cunningham MR. Evaluation of closed incision management with negative pressure wound therapy (CIM): hematoma/seroma and involvement of the lymphatic system. Wound Repair Regen. 2011 Sep-Oct;19(5):588-96. doi: 10.1111/j.1524-475X.2011.00714.x. PMID 22092797
- [Background] Malmsjo M, Huddleston E, Martin R. Biological effects of a disposable, canisterless negative pressure wound therapy system. Eplasty. 2014 Apr 2;14:e15. eCollection 2014. PMID 24741386